CLINICAL TRIAL: NCT07132697
Title: The Efficacy of Intravenous Amino Acids in Reducing the Occurrence of AKI After Live Donor Liver Transplant: An Open Label Randomized Trial
Brief Title: The Efficacy of Intravenous Amino Acids in Reducing the Occurrence of AKI After Live Donor Liver Transplant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEC/2025/119/MA05
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant; Complications; AKI - Acute Kidney Injury
Keywords: Liver Transplantation, Acute Kidney Injury, Amino Acids, KDIGO, NGAL, Randomized Controlled Trial
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino acid mixture infusion with standard of care (Experimental): Continuous infusion of a L-amino acids mixture in a dose of 2 g/kg dry body weight/day (to a maximum 100 g/day) after induction of anesthesia and insertion of CVP line till 72 hours after treatment initiation
  Interventions: Drug: L-Amino acid mixture; Other: Standard of care
- Standard care (Active Comparator): Standard peri liver transplant care as per our institution
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: L-Amino acid mixture — Continuous infusion of a L-amino acids mixture in a dose of 2 g/kg dry body weight/day (to a maximum 100 g/day) after induction of anesthesia and insertion of CVP line till 72 hours after treatment initiation
  Arms: Amino acid mixture infusion with standard of care
Other: Standard of care — Standard peri tranplant care as per out institution including intra operative and post operative care. Its includes starting of immunosuppression after serial blood investigation monitoring.

SUMMARY:
This prospective, open-label, randomized controlled trial aims to evaluate the efficacy of intravenous amino acid infusion in reducing AKI after LDLT. Eligible adult patients undergoing LDLT will be randomized into two groups: one receiving Continuous infusion of a L-amino acids mixture in a dose of 2 g/kg dry body weight/day (to a maximum 100 g/day) after induction of anesthesia and insertion of CVP line till 72 hours after treatment initiation, and the other receiving standard management. The primary outcome is the incidence of AKI as per KDIGO criteria within 7 days of transplant.

DETAILED DESCRIPTION:
This prospective, open-label, randomized controlled trial aims to evaluate the efficacy of intravenous amino acid infusion in reducing AKI after LDLT. Eligible adult patients undergoing LDLT will be randomized into two groups: one receiving Continuous infusion of a L-amino acids mixture in a dose of 2 g/kg dry body weight/day (to a maximum 100 g/day) after induction of anesthesia and insertion of CVP line till 72 hours after treatment initiation, and the other receiving standard management. The primary outcome is the incidence of AKI as per KDIGO criteria within 7 days of transplant.

ELIGIBILITY:
Inclusion Criteria

1. All LDLT Recipient
2. Age: > 18 years
3. Signed informed consent

Exclusion Criteria

1. Negative consent.
2. Pediatric LDLT.
3. ALF patient undergoing LDLT.
4. Patients on intermittent or continuous renal replacement therapy.
5. Patients with eGFR less then 40 ml per min per 1.73 m2.
6. SLKT and prior Kidney transplant.
7. Patient has a hypersensitivity (known allergy) to one or more of the included amino acids.
8. Patient has a known congenital alteration of amino acid metabolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of early post transplant AKI | Within 7 days post transplant
  To compare the incidence of early post transplant AKI (within 1st week) in patients undergoing LDLT between L-amino acids infusion and standard treatment groups

SECONDARY OUTCOMES:
To Determine the severity of early post Liver transplant AKI | 7 days
  To Determine the severity of early post Liver transplant AKI
To determine eGFR at Day 30 and 90. | 90 days
  To determine eGFR at Day 30 and 90.
The use and duration of kidney-replacement therapy during the hospital stay The use and duration of kidney-replacement therapy during the hospital stay | 1 month
  The use and duration of kidney-replacement therapy during the hospital stay The use and duration of kidney-replacement therapy during the hospital stay
The duration of mechanical ventilation, ICU stay and in hospital stay. | 1 month
  The duration of mechanical ventilation, ICU stay and in hospital stay.
In Hospital Mortality | 1 month
  In Hospital Mortality
Major Morbidity (Clavien-Dindo ≥3) and Early Graft Dysfunction. | 1 month
  Major Morbidity (Clavien-Dindo ≥3) and Early Graft Dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ilbs Hospital, D1 Vasant Kunj, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided